CLINICAL TRIAL: NCT06048380
Title: The Effects of Ripasudil in Patients With Fuchs Endothelial Corneal Dystrophy Undergoing Femtosecond Laser Assisted Cataract Surgery
Brief Title: The Effects of Ripasudil in Patients With FED Undergoing Femtosecond Laser Assisted Cataract Surgery
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Singapore Eye Research Institute (Other)
Responsible Party: Principal Investigator, Marcus Ang Han Nian, A/Professor, Singapore Eye Research Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: R1958/01/2023
Record Dates: First submitted 2023-06-26; First posted 2023-09-21 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Fuchs' Endothelial Dystrophy; Cataract
Keywords: Ripasudil
MeSH Terms: conditions — Fuchs' Endothelial Dystrophy; Cataract | interventions — K-115

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment (Experimental): Participants in this group will be asked to instill Glanatec Ophthalmic Solution (containing Ripasadil 0.4%) 4 times a day for 1 month following cataract removal surgery.
  Interventions: Drug: Ripasudil
- Placebo (Placebo Comparator): Participants in this group will be asked to instill saline solution 4 times a day for 1 month following cataract removal surgery.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Ripasudil — Glanatec Ophthalmic Solution 0.4% W/V with ripasudil hydrochloride hydrate as active ingredient is currently being used by patients with ocular hypertension or open-angle glaucoma.
  Inhibition of Rho kinase to facilitate aqueous outflow from the conventional outflow pathway via the trabecular meshwork and Schlemm's canal has been suggested as the IOP-lowering mechanism of action by ripasudil.
  Other Names: Glanatec
  Arms: Treatment
Other: Placebo — Saline eye drops
  Arms: Placebo

SUMMARY:
The purpose of this research is to investigate the effects of ripasudil administered as an ophthalmic solution in patients with FED after femtosecond laser assisted cataract surgery. The secondary aim is to identity the characteristics of patients who will benefit the most with the use of ripasudil based on the test results obtained from this study.

DETAILED DESCRIPTION:
Patients with Fuch's Corneal Endothelial Dystrophy and undergoing femtosecond laser-assisted cataract surgery will be recruited for this study. They will be randomly assigned into treatment or placebo group.

The investigators hypothesize that the ROCK inhibitor ripasudil 0.4% helps maintain corneal endothelial functional integrity and reduce cell loss after cataract surgery in patients with FED.

To test the hypothesis, the investigators plan to conduct a randomized clinical trial which aims to:

1. Evaluate the clinical outcomes of FED eyes following FLACS with and without ripasudil 0.4%
2. To identity which FED patients will most likely benefit from the use of ripasudil 0.4% based on pre-operative parameters
3. To monitor for any adverse effects in patients assigned to ripasudil 0.4%

ELIGIBILITY:
Inclusion Criteria:

1. Patients with FED who will be listed for cataract surgery as part of standard clinical practice (A cataract will be defined as clouding of the lens that interferes with normal vision).
2. Only patients older than 50 years will be included, as cataracts develops with increasing age. No gender criteria are applied.
3. Ability to provide informed consent, and are willing and able to sign a written Informed Consent Form prior to any study-specific procedures.
4. Patients must be willing and able to return for scheduled follow-up examinations for up to 12 months after the surgery.

Exclusion Criteria:

1. Patients who are unable to give consent.
2. An only-functioning eye in a patient who has lost visual potential in the contralateral eye.
3. Diagnosis of clinically relevant eye diseases that may interfere with the aim of the study.
4. History of ripasudil use, as well as other systemic disease such as cardiovascular or renal disease.
5. Patients who have previous allergic reactions to the contents present in Glanatec Ophthalmic solution 0.4%

Ages: 50 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Average endothelial cell density (ECD) is higher in participants in treatment group than participants in placebo. | 3 months
  The ECD at 15 different locations of the cornea is measured with a widefield specular microscope.
  This assessment will be done pre-surgery, Week 1, Week 2, Week 3, 1 month, 3 months post-surgery.

SECONDARY OUTCOMES:
To monitor for conjunctival hyperemia in participants in treatment group. | 3 months
  The Cornea and Contact Lens Research Unit (CCLRU) grading scale will be used as an objective assessment guideline for grading conjunctival hyperaemia.
  The investigators will grade the conjunctival hyperemia This assessment will be done pre-surgery, Week 1, Week 2, Week 3, 1 month, 3 months post-surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Marcus Ang, Principal Investigator — Singapore Eye Research Institute
Locations (1):
- Singapore National Eye Centre, Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No